CLINICAL TRIAL: NCT06192082
Title: Clinical Study About Impacts of Anesthesia Methods on Adverse Cardiovascular Events During Painless Gastroscopy Diagnosis and Treatment in Elderly Frail Patients
Brief Title: Adverse Cardiovascular Events During Painless Gastroscopy Diagnosis and Treatment in Elderly Frail Patients
Acronym: frail
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: frail patients
Record Dates: First submitted 2023-11-27; First posted 2024-01-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia
Keywords: gastroscopy; frail patients; adverse cardiovascular events

STUDY DESIGN:
Intervention Model Description: Using a stratified randomization method, the candidate subjects were divided into two groups: the conscious sedation group (Group A); Intravenous general anesthesia group (Group B); There are 113 cases in each group, with a total of 226 cases in both groups. The computer generated random group numbers will be printed and placed in a separate sealed envelope. When accepting subjects who meet the inclusion criteria, the anesthesiologist will assign the newly recruited subjects to the corresponding groups based on the number in the envelope, and the anesthesiologist will be responsible for recording the physiological characteristics of the patients. Another anesthesiologist followed up the patient after the surgery. Both the follow-up doctor and the patient are unaware of the treatment plan. In emergency situations, anesthesiologists can change the anesthesia method to ensure clinical safety and truthfully record it.
Who Masked: Investigator, Outcomes Assessor
Masking Description: On the premise of ensuring clinical work and safety, in order to objectively evaluate the research results, the single blind method is reasonably used in this project. Patients are unaware of the anesthesia plan, and preoperative data collection and implementation of the anesthesia plan are carried out by experienced anesthesiologists who have undergone detailed training. Postoperative PACU clinical data and postoperative follow-up were followed up by another anesthesiologist who was unaware of the trial group over the phone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The conscious sedation group (Experimental): conscious sedation
  Interventions: Procedure: The conscious sedation group
- Intravenous general anesthesia group (Active Comparator): Intravenous general anesthesia
  Interventions: Procedure: Intravenous general anesthesia group

INTERVENTIONS:
Procedure: The conscious sedation group — The conscious sedation group (Group A) received sufentanil 0.05-0.1 5 minutes before examination μ G/kg, administration time 30 seconds, 1-2 mg of midazolam administered 2 minutes before examination; Evaluate the patient's MOAA/S score, insert a digestive endoscope at 2-3 minutes, and add 1-2mg of midazolam if the patient is unable to tolerate coughing or movement during the examination. Reevaluate the MOAA/S score, and continue the operation after 2-3 minutes;
  Other Names: Group A
  Arms: The conscious sedation group
Procedure: Intravenous general anesthesia group — Intravenous general anesthesia group (Group B): sufentanil 0.05-0.1 μ G/kg, administration time 30 seconds, 1mg/kg of propofol administered 2 minutes before examination. Depending on the patient's sleep status, 10mg of propofol can be administered every 30 seconds; Evaluate the patient's MOAA/S score. At 0-1 points, a digestive endoscope is inserted. If there is coughing or physical activity during the examination that the patient cannot tolerate, propofol 10-20mg can be administered multiple times. Evaluate the MOAA/S score again, and continue the operation after 0-1 points.
  Other Names: Group B
  Arms: Intravenous general anesthesia group

SUMMARY:
This study aims to compare the effects of conscious sedation and intravenous general anesthesia on cardiovascular events in frail patients undergoing digestive endoscopy diagnosis and treatment.

DETAILED DESCRIPTION:
This study aims to compare the effects of conscious sedation and intravenous general anesthesia on cardiovascular events in frail patients undergoing digestive endoscopy diagnosis and treatment.

Both sets of anesthesia plans completed preoperative evaluations, including blood count, coagulation function, liver and kidney function, and cardiopulmonary function. Routine monitoring of electrocardiograms (ECG), non-invasive blood pressure (NIBP), pulse oximetry (SpO2), open veins, and administration of a balance solution of 3-5ml/kg. h. The conscious sedation group (Group A) received sufentanil 0.05-0.1 5 minutes before examination μ G/kg, administration time 30 seconds, 1-2 mg of midazolam administered 2 minutes before examination; Evaluate the patient's MOAA/S score, insert a digestive endoscope at 2-3 minutes, and add 1-2mg of midazolam if the patient is unable to tolerate coughing or movement during the examination. Reevaluate the MOAA/S score, and continue the operation after 2-3 minutes; Intravenous general anesthesia group (Group B): sufentanil 0.05-0.1 μ G/kg, administration time 30 seconds, 1mg/kg of propofol administered 2 minutes before examination. Depending on the patient's sleep status, 10mg of propofol can be administered every 30 seconds; Evaluate the patient's MOAA/S score. At 0-1 points, a digestive endoscope is inserted. If there is coughing or physical activity during the examination that the patient cannot tolerate, propofol 10-20mg can be administered multiple times. Evaluate the MOAA/S score again, and continue the operation after 0-1 points. All anesthetics should be discontinued before the end of the surgery. Since the examination, blood pressure should be measured every 2 minutes, while HR, SpO2, and RR should be recorded to observe if there are any abnormalities in the electrocardiogram. If there are any abnormalities, please explain until the endoscope is removed from the dental pad. Record the satisfaction of gastroenterologists, anesthesiologists, and patients after surgery. Follow up patients by phone within three days after surgery to determine the incidence of adverse events (dizziness, headache, palpitations, wheezing, mobility, nausea and vomiting).

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 65 years old, regardless of gender
2. ASA is classified as Class II and III;
3. BMI 18-28 kg/m2;
4. Patients undergoing examination or treatment outside the operating room;
5. FRAIL scale score ≥ 3 points 6 The patient voluntarily participated in this study and signed an informed consent form.

Exclusion Criteria:

1 Those who are allergic or contraindicated to drugs such as benzodiazepines, opioids, propofol, and their drug components;

2. Acute heart failure; Unstable angina pectoris; Myocardial infarction occurred within 6 months prior to screening; Resting electrocardiogram heart rate<50 beats/minute; Third degree atrioventricular transmission delay; Severe arrhythmia; Moderate to severe heart valve disease;

3. Patients with severe respiratory diseases (acute respiratory infections, acute exacerbations of chronic obstructive pulmonary disease, uncontrolled asthma, etc.);

4. Patients who have not received formal antihypertensive treatment or have poor blood pressure control;

5. Patients with traumatic brain injury, possible presence of intracranial hypertension, cerebral aneurysms, history of cerebrovascular accidents, and central nervous system diseases;

6. Individuals with mental system diseases (schizophrenia, mania, bipolar disorder, mental disorder, etc.), long-term history of taking psychotropic drugs, and cognitive impairment;

7. Other situations that have been determined by the researcher to be unsuitable for inclusion.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Adverse cardiovascular events | during the examination and recovery room time(up to 2 hours)
  The occurrence rate of heart rate abnormal events (defined as heart rate abnormal events with a baseline fluctuation of ± 30%)；The incidence of blood pressure fluctuation events (defined as blood pressure fluctuation events with a baseline blood pressure fluctuation of ± 30%);The incidence of angina, myocardial infarction, cardiac arrest, acute heart

SECONDARY OUTCOMES:
The incidence of other adverse events | during the examination and recovery room time(up to 2 hours)
  The incidence of other adverse events (SPO2<90%, apnea, physical activity, pain, coughing, aspiration, muscle tremor, nausea and vomiting, difficulty breathing, etc.)
VAS score | during the examination and recovery room time(up to 2 hours)
  VAS score, also known as visual simulation score, can be divided into 10 equal parts, with 0 being no pain and 10 being the most painful.
Satisfaction score | during the examination and recovery room time(up to 2 hours)
  Satisfaction of patients, endoscopists, and anesthesiologists.The can be divided into 10 equal parts, with 0 being no satisfaction and 10 being the most satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No